CLINICAL TRIAL: NCT00033943
Title: A Multi-Center, Placebo-Controlled Evaluation of the Safety and Efficacy of Two Dosage Levels of OP2000 (75 Mg and 125 Mg) Administered Once Daily by Subcutaneous Injection for the Treatment of Active Ulcerative Colitis
Brief Title: Safety and Efficacy of OP2000 (Deligoparin) in the Treatment of Active Ulcerative Colitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Incara Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OP201
Record Dates: First submitted 2002-04-16; First posted 2002-04-17 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-10

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

INTERVENTIONS:
Drug: deligoparin

SUMMARY:
This study will evaluate the effectiveness and safety of the experimental compound OP2000 (deligoparin) in patients with active ulcerative colitis. Patients eligible for this study will have received (and will continue to receive) stable doses of aminosalicylates (oral, enema and/or suppository), if tolerated. OP2000 is an ultra low molecular weight heparin with anticoagulant (blood thinning) and anti-inflammatory actions that may be of benefit for the treatment of ulcerative colitis.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, research study to evaluate the effectiveness and safety of the experimental compound OP2000 (deligoparin) in patients with active ulcerative colitis. Patients eligible for this study will have received (and will continue to receive) stable doses of aminosalicylates (oral, enema and/or suppository), if tolerated. OP2000 is an ultra low molecular weight heparin with anticoagulant (blood thinning) and anti-inflammatory actions that may be of benefit for the treatment of ulcerative colitis. Patients will be randomized (assigned by chance like the toss of a coin) to receive 75 mg OP2000, 125 mg OP2000, or placebo once daily for 6 weeks. Study drug will be administered by subcutaneous (under the skin) injection and patients will be taught how to self-administer these injections. Following an initial Screening Visit, eligible patients will return to the clinic for initiation of study treatment and then again for follow-up visits after 1, 2, 4 and 6 weeks of treatment. A follow-up telephone call will be scheduled 2 months (and possibly also 4 and 6 months) after completing study treatment. Study procedures will include a flexible sigmoidoscopy at the Screening Visit and at the Week 6 visit.

ELIGIBILITY:
Inclusion Criteria:

* History of ulcerative colitis at least 3 months with biopsy and colonoscopy confirmation.
* Treatment with aminosalicylates at least 28 days, if tolerated.
* Duration of current flare-up at least 7 days.
* Must be able to self administer once-daily subcutaneous (under the skin) injections of study drug.

Exclusion Criteria:

* Disease limited to the rectum.
* Toxic megacolon.
* The use of anticoagulant drugs.
* A history of any bleeding disorder.
* A history of heparin-induced thrombocytopenia.
* Evidence of liver or kidney impairment.
* Women who are pregnant or breast feeding.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 270
Dates: Start 2001-01; Study Completion 2002-09

CONTACTS AND LOCATIONS:
Locations (33):
- United States (33):
  - AGMG Clinical Research, Anaheim, California
  - Community Clinical Trials, Orange, California
  - Rocky Mountain Gastroenterology Associates, Lakewood, Colorado
  - Rocky Mountain Clinical Research, Littleton, Colorado
  - University of Florida Gainesville/Gainesville VAMC, Gainesville, Florida
  - Borland-Groover Clinic, Jacksonville, Florida
  - University of Miami, Division of Clinical Pharmacology, Miami, Florida
  - Miami Research Associates, Miami, Florida
  - Atlanta Gastroenterology Associates, LLC, Atlanta, Georgia
  - Univ. of Kentucky Medical Center, Lexington, Kentucky
  - Metropolitan Gastroenterology Group, Chevy Chase, Maryland
  - University of Michigan Health System, Ann Arbor, Michigan
  - Minnesota Clinical Research Center, Saint Paul, Minnesota
  - Washington Univ. School of Medicine, St Louis, Missouri
  - Gastroenterology Specialties, PC, Lincoln, Nebraska
  - Long Island Clinical Research Associates, Great Neck, New York
  - Daniel H. Present, MD, New York, New York
  - Univ. of North Carolina Hospital, Chapel Hill, North Carolina
  - Charlotte Gastroenterology & Hepatology, PLLC, Charlotte, North Carolina
  - Duke Health Center, Durham, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Consultants for Clinical Research, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oklahoma Foundation for Digestive Research, Oklahoma City, Oklahoma
  - Gastroenterology United of Tulsa, Tulsa, Oklahoma
  - West Hills Gastroenterology, Portland, Oregon
  - Hospital of the Univ. of Pennsylvania, Philadelphia, Pennsylvania
  - Memphis Gastroenterology Group, PC, Memphis, Tennessee
  - Nashville Clinical Research, Nashville, Tennessee
  - GANT Research, PA, Fort Worth, Texas
  - Gastroenterology Clinic of San Antonio, San Antonio, Texas
  - Univ. of Virginia Health System, Charlottesville, Virginia
  - Wisconsin Center for Advanced Research, LLC, Milwaukee, Wisconsin